CLINICAL TRIAL: NCT04302610
Title: The Use of a Heat and Moisture Exchange Mask to Reduce Exercise Induced Bronchoconstriction Severity and Improve the Airway Health of Individuals With Asthma
Brief Title: Do Heat and Moisture Exchange Mask Reduce EIB and Cough Severity in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kent (Other)
Collaborators: Asthma UK (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AUK-IG-2016-332
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2016-05

CONDITIONS: Asthma, Exercise-Induced; Asthma
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma

STUDY DESIGN:
Intervention Model Description: randomised cross-over design
Who Masked: Participant
Masking Description: Heat Exchange Mask SHAM Mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HME MASK (Experimental): During the Exercise, participants wore either an HME mask (MASK) (ColdAvenger® expedition balaclava, USA, www.coldavenger.com)
  Interventions: Device: Heat and Moisture Exchange mask (ColdAvenger® expedition balaclava, USA,
- SHAM mask (Sham Comparator): a sham mask (SHAM) which was the same HME mask with holes cut across the entire ventilator cup and the ventilator removed
  Interventions: Device: Sham treatment
- Control (No Intervention): No mask (CONT) wearing only the balaclava to which the HME and SHAM mask were attached. Mouth and face not covered.

INTERVENTIONS:
Device: Heat and Moisture Exchange mask (ColdAvenger® expedition balaclava, USA, — A heat and moisture exchange mask will warm and humidify inspired air and therefore reduce airway heat and water loss during exercise. This will potentially reduce the incidence of and severity of EIB and may also have the potential to decrease the incidence of cough amongst athletes engaging in sports in cold dry environments
  Arms: HME MASK
Device: Sham treatment — Same as the HME mask but active HME parts withdrawn from devices and multiple holes made in mouth piece to improve ventilation of mask and reduce HME ability of mask
  Arms: SHAM mask

SUMMARY:
The overall aim of this study is to determine if face masks that can warm and humidify air can improve overall asthma control and markers of airway health during exercise in cold dry environments. We will investigate the potential protective benefits of the face masks against exercise induced asthma during 1) a "one-off" bout of exercise in a cold dry environment and 2) over the course of a four week period, exercising three times per week in a cold dry environment.

DETAILED DESCRIPTION:
Physical activity is recognised as a trigger for individuals with asthma, however regular physical activity is considered to be important in the overall management of the condition. There is clear evidence that demonstrates if individuals with asthma engage with regular physical activity they will improve their physical fitness and breathing control, whilst at the same time experiencing reductions in asthma severity, symptoms, and medication use. In addition undertaking regular exercise reduces the risk of developing other diseases such as heart disease or type 2 diabetes. Despite the clear health benefits of engaging in regular physical activity there is evidence that some people with asthma avoid physical activity due to shortness of breath, worsening asthma symptoms during physical activity or fear of experiencing such symptoms.

Physical activity in cold dry environments exacerbates symptoms for many individuals with asthma resulting in greater avoidance of physical activity during the winter months. The increased risk of asthma from exercising in cold environments has led to Asthma UK advising susceptible individuals to avoid exercise outside in cold environments (http://www.asthma.org.uk/advice-exercise). This places obvious constraints and limitations on individuals with asthma for whom the aim of optimum treatment is to allow them to follow a "normal" lifestyle. Indeed, exposure to cold air on exertion is relevant to a significant proportion of individuals with asthma who engage with outdoor physical activity as part of their daily routine; e.g. cycle-commuting to work, outdoor construction workers.

A mask that is able to warm and humidify the air during exercise may provide a solution for asthmatic individuals susceptible to cold dry environments. There are a limited number of small studies that provide tentative evidence suggesting masks which warm and humidify air can protect against reductions in lung function during and following physical activity. However, it is unknown whether the use of these masks provides protection against the mechanisms that drive asthmatic symptoms. It is also unclear whether using the masks over a prolonged period of time significantly reduces asthma severity, inhaler use, or presence of symptoms.

The overall aim of this study is to determine if face masks that can warm and humidify air can improve overall asthma control and markers of airway health during exercise in cold dry environments. We will investigate the potential protective benefits of the face masks against exercise induced asthma during 1) a "one-off" bout of exercise in a cold dry environment and 2) over the course of a four week period, exercising three times per week in a cold dry environme

ELIGIBILITY:
Inclusion Criteria:

* Ability to consent to the research
* Prior clinician based diagnosis of asthma
* Males and females
* 18 - 45 years
* Engage in regular exercise (at least twice weekly)
* Normal resting Forced Expiratory Volume in One Second (FEV1); defined as greater than 80% of predicted value.

Exclusion Criteria:

* Chest infection within the past 4 weeks, or any other illness within the past 2 weeks
* Fall in FEV1 >50% from baseline following exercise challenge (see protocol)
* Baseline FEV1 of < 80% of predicted
* Cardiovascular conditions:

  * Coronary Artery Disease
  * High Blood Pressure
  * Heart Failure
  * Diagnosed Abnormality of Heart Rhythm
* Metabolic diseases:

  * Type 1 diabetes
  * Type 2 diabetes
  * Pre-diabetes
* Daily use of oral corticosteroids
* Hospitalisation due to asthma in the six months prior to study commencement
* Injury or conditions that limit mobility
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
% fall in FEV1 | 30 minutes
  Change in Forced Expiratory Volume in One Second from baseline to post exercise

SECONDARY OUTCOMES:
coughs per hour after EX | 24 hours
  Number of coughs per hour in a 24 hour period after exercise

CONTACTS AND LOCATIONS:
Overall Officials: John W Dickinson, PhD, Principal Investigator — University of Kent

IPD SHARING:
Plan to Share IPD: No